CLINICAL TRIAL: NCT03505151
Title: Absolute Bioavailability and Pharmacokinetics of BI 409306 Using a Single Oral Dose of BI 409306 Co-administered With an Intravenous Stable Labeled Isotope BI 409306 (C-13/N-15) in Healthy Male and Female Subjects (Non-Randomised, Open-label, Single Arm, Single Period Design)
Brief Title: This Study in Healthy Men and Women Tests How the Body Takes up BI 409306
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1289-0025; 2017-004798-14 (EudraCT Number)
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — BI 409306

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BI 409306 tablet + intravenous isotope BI 409306 (C-13/N-15) (Experimental): On day 1, subjects were administered the Test treatment (T): a single dose of 50 milligram (mg) of BI 409306 film-coated tablet orally with 240 milliliter (mL) of water, followed 30 minutes (min) later by the Reference treatment (R): 0.1 mg isotope BI 409306 (C-13/N-15) as intravenous (i.v.) infusion over 30 minutes.
  Both treatments were given in fasted state.
  Interventions: Drug: BI 409306 (C-13/N-15); Drug: BI 409306

INTERVENTIONS:
Drug: BI 409306 (C-13/N-15) — i.v solution
Drug: BI 409306 — Film-coated tablet

SUMMARY:
The primary objective of this trial is to investigate the absolute bioavailability of BI 409306. The secondary objective is the evaluation and comparison of several pharmacokinetic parameters for the different treatments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 55 years (incl.)
* BMI of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation
* Known CYP 2C19 metabolizer status
* Male subjects, or female subjects who meet any of the following criteria starting from at least 30 days before the first administration of trial medication and until 30 days after trial completion:

  * Use of adequate contraception, e.g. non-hormonal intrauterine device plus condom.
  * Sexually abstinent
  * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
  * Surgically sterilised (including hysterectomy)
  * Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of FSH (follicle stimulating hormone) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Current smoker or ex-smoker who quit smoking less than 30 days prior to screening
* Alcohol abuse (consumption of more than 20 g per day for females and 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 msec in males or repeatedly greater than 470 msec in females) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

Female subjects will not be allowed to participate if any of the following applies:

* Positive pregnancy test, pregnancy or plans to become pregnant within 30 days after study completion
* Lactation period
* Concomitant use of hormonal replacement therapy or hormonal contraceptives

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2018-05-19 (Actual); Study Completion 2018-05-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was a non-randomized, open-label, single arm, single period, phase 1 clinical trial in healthy subjects in order to compare the reference treatment (R) which consisted of an infusion of 0.1 mg intravenously administered stable labeled isotope BI 409306 (C-13/N-15); with 50 mg of orally administered unlabeled BI 409306 (Test treatment, T).
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist sites to ensure that they (the subjects) met all implemented inclusion/exclusion criteria. Subjects were not to be entered to trial drug if any of the specific entry criteria was violated.
Period: Overall Study
Arm/Group | BI 409306 Tablet + Intravenous Isotope BI 409306 (C-13/N-15)
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The TS included all subjects who were documented to have taken at least one dose of trial medication.
Arm/Group | BI 409306 Tablet + Intravenous Isotope BI 409306 (C-13/N-15)
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.8 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 409306 and Stable Labelled Isotope BI 409306 (C-13/N-15) Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 409306 and stable labelled isotope BI 409306 (C-13/N-15) over the time interval from 0 extrapolated to infinity (AUC0-∞). The dose-normalized values for AUC0-∞ are reported.
Time Frame: T and R:Within 3 hours (h) before dosing, 0.75h, 0.97h, 1.333h, 1.75h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 7h, 8h, 9h, 10h, 12h and 24h after dosing. Only T: 0.17h, 0.333h, 0.47h. Only R:0.58h, 0.83h, 1.17h, 1.5h.
Population: Pharmacokinetic Set (PKS). The PKS included all subjects from the TS who provided at least 1 primary PK parameter that was not excluded due to a protocol violation relevant to the evaluation of PK or due to non-evaluability.
Measure: Least Squares Mean (Standard Error); unit: millimole*hour/L/kg [mmol*h/L/kg]
Groups:
- Test Treatment (T): BI 409306; Reference Treatment (R): BI 409306 C-13/N-15: On day 1, subjects were administered the Test treatment (T): a single dose of 50 milligram (mg) of BI 409306 film-coated tablet orally with 240 milliliter (mL) of water, followed 30 minutes (min) later by the Reference treatment (R): 0.1 mg isotope BI 409306 (C-13/N-15) as intravenous (i.v.) infusion over 30 minutes.
  Both treatments were given in fasted state.
Arm/Group | Test Treatment (T): BI 409306 | Reference Treatment (R): BI 409306 C-13/N-15
Number analyzed (Participants) | 9 | 9
millimole*hour/L/kg [mmol*h/L/kg] | NA (NA) — Least squares mean is actually adjusted geometric mean (gMean). Adjusted geometric mean (gMean)= 28.41 Standard error is actually geometric standard error. Geometric standard error = 1.20 | NA (NA) — Least squares mean is actually adjusted geometric mean (gMean). Adjusted geometric mean (gMean)= 63.66 Standard error is actually geometric standard error. Geometric standard error = 1.20
Statistical Analysis 1: Comparison: Test Treatment (T): BI 409306 vs Reference Treatment (R): BI 409306 C-13/N-15; Absolute bioavailability was evaluated using an Analysis of variance model (ANOVA) on BI 409306 AUC0-inf versus 0.1 mg BI 409306 C-13/N-15 i.v. This model included effects accounting for the following sources of variation: 'subjects' and 'formulation'. The effect 'subjects' was considered as random, whereas 'formulation' was considered as fixed. The dose normalised PK endpoints were log transformed (natural logarithm) prior to fitting the ANOVA model; Test type: Other; Ratio T/R = 44.63, 90% CI [32.62 to 61.06], Standard Error of Mean 36.9 — Standard Error of the mean is actually Intra-individual geometric coefficient of variation (gCV) of the mean

2. Primary Outcome: Maximum Measured Concentration of BI 409306 and Stable Labelled Isotope BI 409306 (C-13/N-15), (Cmax)
Description: Maximum measured concentration of the analyte BI 409306 and stable labelled isotope BI 409306 (C-13/N-15), (Cmax).
  The dose-normalized values for Cmax are reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: picomole/Liter/microgram [pmol/L/μg]
Arm/Group | Test Treatment (T): BI 409306 | Reference Treatment (R): BI 409306 C-13/N-15
Number analyzed (Participants) | 9 | 9
picomole/Liter/microgram [pmol/L/μg] | NA (NA) — Least squares mean is actually adjusted geometric mean (gMean). Adjusted geometric mean (gMean)= 23.45 Standard error is actually geometric standard error. Geometric standard error = 1.25 | NA (NA) — Least squares mean is actually adjusted geometric mean (gMean). Adjusted geometric mean (gMean)= 49.63 Standard error is actually geometric standard error. Geometric standard error = 1.25
Statistical Analysis 1: Comparison: Test Treatment (T): BI 409306 vs Reference Treatment (R): BI 409306 C-13/N-15; Ratios of BI 409306 for Cmax versus 0.1 mg BI 409306 C-13/N-15 i.v. was evaluated using ANOVA model. This model included effects accounting for the following sources of variation: 'subjects' and 'formulation'. The effect 'subjects' was considered as random, whereas 'formulation' was considered as fixed. The dose normalised PK endpoints were log transformed (natural logarithm) prior to fitting the ANOVA model; Test type: Other; Ratio T/R = 47.25, 90% CI [27.38 to 81.55], Standard Error of Mean 68.8 — Standard Error of the mean is actually Intra-individual geometric coefficient of variation (gCV) of the mean

3. Secondary Outcome: Terminal Half-life of BI 409306 and Stable Labelled Isotope BI 409306 (C-13/N-15) in Plasma (t1/2)
Description: Terminal half-life of BI 409306 and stable labelled isotope BI 409306 (C-13/N-15) in plasma (t1/2) is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)
Arm/Group | Test Treatment (T): BI 409306 | Reference Treatment (R): BI 409306 C-13/N-15
Number analyzed (Participants) | 9 | 9
hour (h) | 1.49 (23.1) | 1.39 (24.3)

4. Secondary Outcome: Time From Dosing to Maximum Measured Concentration of BI 409306 and Stable Labelled Isotope BI 409306 (C-13/N-15) in Plasma (Tmax)
Description: Time from dosing to maximum measured concentration of BI 409306 and stable labelled isotope BI 409306 (C-13/N-15) in plasma is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Test Treatment (T): BI 409306 | Reference Treatment (R): BI 409306 C-13/N-15
Number analyzed (Participants) | 9 | 9
hour (h) | 0.333 [0.333 to 1.75] | 0.467 [0.333 to 0.467]

5. Secondary Outcome: For: BI 409306 (C-13/N-15): Total Clearance (CL) of BI 409306 (C-13/N-15)
Description: Total clearance (CL) of BI 409306 (C-13/N-15) is reported.
Time Frame: Within 3 hours (h) before drug administration, 0.58h, 0.75h, 0.83h, 0.97h, 1.17h, 1.333h, 1.5h, 1.75h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 7h, 8h, 9h, 10h, 12h and 24h after dosing.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter/minute (mL/min)
Arm/Group | Reference Treatment (R): BI 409306 C-13/N-15
Number analyzed (Participants) | 9
milliliter/minute (mL/min) | 825 (33.6)

6. Secondary Outcome: For BI 409306 (C-13/N-15): Apparent Volume of Distribution During the Terminal Phase After Intravascular Administration (Vz) of BI 409306 (C-13/N-15)
Description: Apparent volume of distribution during the terminal phase after intravascular administration of BI 409306 (C-13/N-15) is reported.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Reference Treatment (R): BI 409306 C-13/N-15
Number analyzed (Participants) | 9
Liter (L) | 98.9 (21.5)

7. Secondary Outcome: Absolute Bioavailability of BI 409306 (Fabs)
Description: The evaluation of the absolute bioavailability (Fabs) of BI 409306 was performed by calculating the ratio between the area under the concentration-time curve over the time interval from 0 extrapolated to infinity (AUC0-∞) determined for the oral treatment (T) and the (AUC0-∞) determined for the i.v. infusion (R), corrected by the respective dose, and multiplied by 100.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: % of bioavailability
Arm/Group | BI 409306 Tablet + Intravenous Isotope BI 409306 (C-13/N-15)
Number analyzed (Participants) | 9
% of bioavailability | 44.6 (54.0)

ADVERSE EVENTS:
Time Frame: From first drug administration until 24 hours after the last oral drug administration, up to 2 days
Description: Treated set (TS): This subject set includes all subjects who were documented to have received at least one dose of study drug.
  The 50 milligram (mg) BI 409306 film-coated tablet, and the 0.1 mg isotope BI 409306 (C-13/N-15) intravenous infusion were administered 30 minutes apart. Therefore, the Adverse Events cannot be assigned to each treatment.
Arm/Group | BI 409306 Tablet + Intravenous Isotope BI 409306 (C-13/N-15)
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 409306 Tablet + Intravenous Isotope BI 409306 (C-13/N-15) (N=9)
Chromatopsia (Eye disorders) | 1
Erythropsia (Eye disorders) | 1
Visual impairment (Eye disorders) | 3

LIMITATIONS AND CAVEATS:
Since no balancing of gender was needed according to the Clinical trial protocol, the use of the volunteers' pool of the trial site, in which male subjects are predominant, resulted in only male subjects being included in this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-05-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT03505151/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT03505151/SAP_001.pdf